CLINICAL TRIAL: NCT04035525
Title: Pharmacokinetic Study on Three Formulations of Coenzyme Q10 With Different Carriers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mélanie Plourde (Other)
Responsible Party: Sponsor-Investigator, Mélanie Plourde, Principal investigator, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MaxSimil and CoQ10
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — coenzyme Q10; Rice Bran Oil

STUDY DESIGN:
Intervention Model Description: Double-blind controlled-randomized pharmacokinetic (PK) study with crossover design (15 men and 15 women), with a minimum of 6 days between treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the research nurse will know the administration order of the different treatments administered. All plasma samples collected during the research project will be anonymized i.e. it will not be possible to identify the participant by his name since a number will be assigned to him. The code key linking the participant's name to his number will be stored, with access restricted to those designated by the principal investigator. The data file is also protected by a password.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MaxSimil® fish oil + CoQ10 (Experimental): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of 1 g MaxSimil® fish oil + 200 mg CoQ10. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: MaxSimil® fish oil + CoQ10
- Rice bran oil + CoQ10 (Active Comparator): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of 1 g rice bran oil + 200 mg CoQ10. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: Rice bran oil + CoQ10
- CoQ10 as powder form (Active Comparator): The participant will arrive fasted at he research center. After installing a cathether and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of 1 g rice bran oil + 200 mg CoQ10. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: CoQ10 as powder form

INTERVENTIONS:
Dietary Supplement: MaxSimil® fish oil + CoQ10 — The intervention is a randomized double blind cross over design testing the pharmacokinetics of 1) CoQ10 combined with MaxSimil fish oil as a carrier, 2) CoQ10 combined with rice bran oil as a carrier, and 3) CoQ10 as a powder form.
  Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours. Each participant will perform all three treatments, with a minimum of 7 days between treatments. A questionnaire will document the side effects felt by participants.
  Arms: MaxSimil® fish oil + CoQ10
Dietary Supplement: Rice bran oil + CoQ10 — The intervention is a randomized double blind cross over design testing the pharmacokinetics of 1) CoQ10 combined with MaxSimil fish oil as a carrier, 2) CoQ10 combined with rice bran oil as a carrier, and 3) CoQ10 as a powder form.
  Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours. Each participant will perform all three treatments, with a minimum of 7 days between treatments. A questionnaire will document the side effects felt by participants.
  Arms: Rice bran oil + CoQ10
Dietary Supplement: CoQ10 as powder form — The intervention is a randomized double blind cross over design testing the pharmacokinetics of 1) CoQ10 combined with MaxSimil fish oil as a carrier, 2) CoQ10 combined with rice bran oil as a carrier, and 3) CoQ10 as a powder form.
  Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours. Each participant will perform all three treatments, with a minimum of 7 days between treatments. A questionnaire will document the side effects felt by participants.
  Arms: CoQ10 as powder form

SUMMARY:
Coenzyme Q10 (CoQ10) is a vitamin-like substance produced in all living human cells and naturally occurring in dietary sources. In addition to being responsible for the synthesis of adenosine triphosphate (ATP), a major source of energy, CoQ10 plays an essential role in maintaining several biochemical pathways of the human body: i) it acts as a primary scavenger of free radicals, and ii) it protects membranes phospholipids from peroxidation and membranes proteins and mitochondrial DNA from oxidative damage. Despite the potential impact that it has shown in a wide array of health conditions, CoQ10 has been reported to have a poor bioavailability in humans with a slow and incomplete absorption from the small intestine. This has been attributed to its high molecular weight, strongly lipophilic nature and low aqueous solubility. To overcome the above limitations, various drug delivery systems such as liposomes, polymeric nanoparticles, polymeric micelles, solid lipid nanoparticles, nanostructured lipid carriers, self-emulsifying systems, nanoemulsions and solid and aqueous dispersions have been explored and developed to improve the solubility, the absorption and the bioavailability of CoQ10. Even though these different technologies and delivery systems were able to improve the absorption of CoQ10 and increase its bioavailability, the carriers used to deliver CoQ10 are based on synthetic products with no health benefits attributed to them. Aligned with its mission and vision to provide its clients with wellness products, Biodroga Neutraceuticals Inc developped a CoQ10 product using its patented MaxSimil technology that is based on omega-3 fatty acids (EPA and DHA) and this health product will be serving as the carrier for CoQ10. Therefore, the aim of this study is to perform a PK study using a powder product of CoQ10 and a rice bran oil + CoQ10 forms as comparators to the MaxSimil® + CoQ10 omega-3 supplement and compare their bioavailability and side effects. In this context, a randomized crossover design with a minimum of 7 days of washout between treatments will be used. The MaxSimil® + CoQ10 formulation is anticipated to provide the best vehicle to increase the bioavailability of CoQ10 with the lowest side effects for the participants.

DETAILED DESCRIPTION:
Benefits and importance of CoQ10 for the human health:

Coenzyme Q10 (CoQ10) is an endogenously produced lipid-soluble molecule of the human organism that is considered an essential component of the mitochondrial electron transport chain where it is the electron acceptor for complexes I and II. In this context, CoQ10 plays a key role in mitochondrial oxidative phosphorylation and ATP production and therefore it is essential for all energy-dependent processes in the body, enhancing the immune-system and acting as a free radical scavenger. In addition to its abundant presence in the mitochondrion, CoQ10 is found in other organelles such as endoplasmic reticulum, peroxisomes, lysosomes and vesicles. It is a membrane stabilizer, preserves myocardial sodium-potassium ATPase activity, and stabilizes myocardial calcium-dependent ion channels. Several factors such as ageing, poor eating habits, stress and infection, are known to affect the organism's ability to continue synthesizing and providing the adequate amounts of CoQ10. With age, the human organism begins to develop a CoQ10 deficiency due to its inability to synthesize it from food where it is present in beef, poultry, broccoli, soya oil and peanuts. In this context, several researchers have advised using CoQ10 supplements alone or in combination with other nutritional supplements to alleviate this deficiency and help maintain health of elderly people or treat some of the health problems or diseases. Due to these functions, CoQ10 finds its application in different commercial branches such as food, cosmetic, or pharmaceutical industries. The antioxidant activity of CoQ10 surpasses both in the amount and in efficiency other antioxidants. The protective effect is extended to lipids proteins and DNA mainly because of its close localization to the oxidative events and the effective regeneration by continuous reduction at all locations. CoQ10 in its reduced form as a hydroquinone (ubiquinol) is a potent lipophilic antioxidant that has a great importance as a free radical scavenger. CoQ10 protects the stability of the cell membranes, protects DNA from free radical induced oxidative damage, and is capable of recycling and regenerating other antioxidants, such as tocopherol and ascorbate. Other important functions of CoQ10 as e.g. cell signaling and gene expression have also been described.

Absorption and Transport of CoQ10:

Taking its lipophilic nature, the absorption of CoQ10 is enhanced in the presence of lipids with the main role attributed to the intestinal secretions from the pancreas and bile that are known to facilitate emulsification and micelle formation required for the fats absorption. Either during or following its absorption in the intestine, CoQ10 is reduced to ubiquinol, incorporated into chylomicrons and then transported via the lymphatics to the circulation where about 95% of CoQ10 in circulation exists in its reduced form as ubiquinol in human subjects. Plasma CoQ10 concentrations are highly dependent on plasma lipoproteins where CoQ10 redistributes possibly to protect lipoproteins from oxidation. Several factors have highlighted the poor absorption of orally administered CoQ10 such as its insolubility in water, limited solubility in lipids, and relatively large molecular weight. A preclinical study has reported that only about 2-3% of orally-administered CoQ10 was absorbed. Additionally, the absorption of CoQ10 and its bioavailability have been shown to be dependent on other factors such as the nature of the formulation of CoQ10 with solubilized formulations been reported to have an advanced effect on the bioavailability.

Tissue distribution of CoQ10 in humans and animals:

Upon its presence in the circulatory system, CoQ10 is distributed in all the tissues in varying amounts with high concentrations been reported to be present in organs with high metabolic activities such as the heart, kidney, liver and muscle. Additionally, and due to its lipophilic nature, the lipid content of the body organ do play a role in the CoQ10 distribution. At the subcellular level, data have shown that a large portion of CoQ10 (40-50%) is localized in the mitochondrial inner membrane, with smaller amounts in the other organelles and in the cytosol. At the blood level, about 95% of CoQ10 is present in the ubiquinol-reduced form. Among blood cells, lymphocytes and platelets contain significant amounts of CoQ10 whereas red blood cells contain only a tiny amount due to their lack of mitochondria.

Pharmacokinetics of CoQ10:

In a pharmacokinetic study conducted on sixteen healthy subjects, and using deuterium-labeled CoQ10 (100 mg), a Tmax of 6.5 h along with an elimination half-life of about 33 hours and a mean plasma levels around 1 µg/ml have been reported. Similar results have been also found when unlabeled CoQ10 has been used in another study. It is worth to mention that powder-based CoQ10 products were used in both of these studies. To compare the bioavailability of several CoQ10 formulations, three different solubilized formulations of CoQ10 were compared to a powder-based formulation. Results have shown that two of the solubilized formulations along with the powder product have showed a Tmax of about 6 h whereas the remaining solubilized formulation had a Tmax of about 8 h. These results were similar and in accordance to other results. The Tmax value of about 6 h or longer indicates that CoQ10 is absorbed slowly from the gastrointestinal tract and this is attributable to both its hydrophobicity and high molecular weight. In the different pharmacokinetic studies conducted on CoQ10, a second plasma CoQ10 peak has been observed at about 24 h following oral ingestion, which may be due to both enterohepatic recycling and redistribution from the liver to circulation.

Bioavailability of CoQ10 / Delivery systems:

Although CoQ10 has been reported to be useful for the treatment of several diseases such as ageing, fatigue, irregular heartbeat, high blood pressure, and immune system impairment among others, its efficacy has been always hindered by its high lipophilicity and poor solubility in water, which leads to decreased absorption into the systemic circulation. Several conventional formulations of CoQ10 are available in the form of soft gel capsules, oral spray and tablets. Despite these, the idea of delivery of CoQ10 to the body remains a challenge. To overcome the slow absorption of CoQ10, various bioavailability enhancement methods have been developed such as liposomes, polymeric nanoparticles, polymeric micelles, solid lipid nanoparticles, nanostructured lipid carriers, self-emulsifying systems, nanoemulsions and solid and aqueous dispersions have been explored and developed to improve the solubility, the absorption and the bioavailability of CoQ106. Based on purified phospholipids as the key component and with a dose of 100 mg of CoQ10, NanoSolve has shown to increase the bioavailability of CoQ10 fivefold in comparison to pure CoQ109. Using cyclodextrin as a carrier, a novel patented formulation known as Q10Vital® has demonstrated its ability to increase the bioavailability of CoQ10 when two Q10Vital formulations (liquid and powder) were compared to regular CoQ10/soybean oil softgels. Although no difference in the Tmax was observed between the three tested products, both Q10Vital formulations have reported a higher Δcmax (32 % for the liquid formulation and 25% for the powder formulation) in comparison with the regular softgel product.

Rationale of this study:

Although several technologies and delivery systems have been used to improve the absorption of CoQ10 and increase its bioavailability, the carriers used to deliver CoQ10 are based on synthetic products with no health benefits attributed to them. In alignment with its mission and vision to deliver wellness products, Biodroga Neutraceuticals Inc has decided to develop a new product (MaxSiQ10) aiming to increase the absorption and the bioavailability of CoQ10 by using omega-3 fatty acids as a vector delivery system and a carrier for CoQ10. The benefits of omega-3 fatty acids to the human health have been well documented and reported in several studies20-22. Because the human body does not efficiently produce fish-derived omega-3 fatty acids (EPA and DHA) from its precursor alpha-linolenic acid, it is necessary to obtain adequate amounts through fish and fish-oil products. Studies have shown that EPA and DHA have been associated with better fetal development, including neuronal, retinal, and immune function. Additionally, EPA and DHA may affect many aspects of cardiovascular function including inflammation, peripheral artery disease, major coronary events, and anticoagulation. Promising results have been attributed for EPA and DHA in weight management, and prevention of cognitive decline. To differentiate themselves from the other products and technologies already existing on the market, Biodroga Neutraceuticals Inc will be using its MaxSimil® technology as the vector delivery system for CoQ10. MaxSimil is a new-patented delivery technology that intrinsically enhances the absorption of omega-3 fatty acids (EPA and DHA) of a given fish oil by modifying its glyceride composition to simulate digestion. This technology delivers "absorption-ready" formulations enriched with "self emulsifing" monoglycerides (MAG) and have the potential to be better absorbed when compared to the more traditional ethyl ester (EE) and reconstituted triglycerides (rTG) fish oil forms available on the market today. What differentiates MaxSimil relies in being a completely natural health product with a demonstrated ability to increase the absorption of omega-3 fatty acids whereas other carriers are synthetic chemical surfactants with detrimental effects on human cells. Therefore, this project will test a MAG-Omega-3 formulation enriched with CoQ10, since it was hypothesized that this formulation will be the most absorbed and bioavailable with the lowest side effects in men and women without any disease such as intestinal lipid absorption issues.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 50 years old (inclusive).
* Body mass index between 18,5 and 34,9 at the selection visit (inclusive).
* Normal to moderately elevated lipidemia (total cholesterol ≤ 240 mg / dl, LDL ≤ 160 mg / dl, TG ≤ 199 mg / dl).
* Woman of child bearing potential must accept to use an effective contraceptive method for the duration of the study.

Exclusion Criteria:

* Tobacco.
* Current or past performance athlete.
* Allergy to fish or seafood.
* Special diet like a fat-free, vegetarian or vegan diet.
* Menopause or pre-menopause with amenorrhea > 6 months.
* History of current or past alcohol and / or drug abuse.
* Pregnant women or nursing women.
* Malnutrition (assessed by albumin, hemoglobin and blood lipid levels).
* Systemic disease: vasculitis, Lupus Erythrocyte Disseminated (SLE), sarcoidosis, cancer (except if in remission for more than 10 years and without cerebral involvement), uncompensated hypothyroidism, vitamin B12 deficiency not supplemented and / or complicated, diabetes, insufficiency severe renal.
* Abnormal liver, kidney or thyroid function; these conditions will not exclude a patient if he / she has been stabilized on treatment for at least 3 months and there has been no recent change in his / her medication.
* Cardiac event or recent major surgery (<6 months).
* Person with a history of thrombosis or haemorrhagic diathesis.
* People who have a malabsorption disease such as pancreatitis, Crohn's disease or who have had bariatric surgery.
* Hypo or hypertension.
* People consuming omega 3 fatty acid supplements for more than 6 months.
* Parkinson disease.
* Down syndrome.
* Known psychiatric history: schizophrenia, psychotic disorders, major affective disorder (bipolar disorder and major depression <5 years), panic disorder, Compulsive Obsessive Compulsive Disorder (OCD).
* Epilepsy, cerebral trauma with loss of consciousness, subarachnoid hemorrhage.
* Medication affecting fat absorption (ie, Orlistat, Alli, etc.), which interferes with the uptake of omega-3 fatty acids (ie, anticoagulants like coumadin, aspirin is not an exclusion criterion (Watson et al, 2009)), which affects lipid metabolism (ie, all types of drugs to lower cholesterol or triglycerides) or which affect CoQ10 blood levels (b-blockers and hypoglycemic agents).
* Person who has donated blood or had significant blood loss in the 30 days prior to the start of the study.
* Not available to perform the 3 different treatments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Determine the bioavailability of CoQ10 in combination with fish oil, rice oil or alone: Calculating the area under the curve (AUC) 0-48h as the first parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours post-treatment.
  Plasma CoQ10 levels will be measured by high-performance liquid chromatography (HPLC), each sample being performed randomly blindly. After HPLC analyzes, area under the curve (AUC) 0-48 hours will be calculated, as the first parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of CoQ10 in combination with fish oil, rice oil or alone: Calculating the AUC 0-6h (absorption study) as the second parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours post-treatment.
  Plasma CoQ10 levels will be measured by high-performance liquid chromatography (HPLC), each sample being performed randomly blindly. After HPLC analyzes, AUC 0-6 hours (absorption study) will be calculated, as the second parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of CoQ10 in combination with fish oil, rice oil or alone: Calculating the maximum concentration as the third parameter of the PK. | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours post-treatment.
  Plasma CoQ10 levels will be measured by high-performance liquid chromatography (HPLC), each sample being performed randomly blindly. After HPLC analyzes, maximum concentration will be calculated, as the third parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of CoQ10 in combination with fish oil, rice oil or alone: Calculating the time when the maximum concentration is reached, as the fourth parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. HPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 4, 5, 6, 8, 10, 12, 24 and 48 hours post-treatment.
  Plasma CoQ10 levels will be measured by high-performance liquid chromatography (HPLC), each sample being performed randomly blindly. After HPLC analyzes, time when the maximum concentration is reached will be calculated, as the fourth parameter of the PK. Statistical analyzes will then be performed on this PK parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada